CLINICAL TRIAL: NCT01504048
Title: Prospective Study on the Usefulness of Chromoendoscopy in Detecting Microscopic Colitis in Patients Undergoing Colonoscopy Due to Chronic Watery Diarrhoea
Brief Title: Usefulness of Chromoendoscopy in Diagnosing Microscopic Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Peter Thelin Schmidt, Head of Endoscopy, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PTS-02
Record Dates: First submitted 2011-12-29; First posted 2012-01-05 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Diarrhoea; Lymphocytic Colitis; Collagenous Colitis
Keywords: Microscopic colitis; Intestinal Diseases; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Lymphocytic; Colitis, Collagenous; Colitis, Microscopic; Intestinal Diseases; Inflammatory Bowel Diseases | interventions — Colonoscopy; Indigo Carmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chromoendoscopy (Experimental)
  Interventions: Procedure: Colonoscopy with Indigo-Carmine Chromoendoscopy

INTERVENTIONS:
Procedure: Colonoscopy with Indigo-Carmine Chromoendoscopy — Colonoscopy with chromoendoscopy using 0.2-0.5% Indigo-Carmine solution sprayed in five areas of the large intestine: Cecum, ascending colon, transverse colon, descending colon and rectum. Pictures are taken before and after dye-spraying and biopsies are collected from all segments of the large intestine and rectum.
  Other Names: Indigo-Carmine

SUMMARY:
The purpose of this study is to determine whether chromoendoscopy using Indigo-Carmine dye spray is useful in diagnosing microscopic colitis among patients undergoing colonoscopy due to chronic watery diarrhea.

DETAILED DESCRIPTION:
Microscopic colitis is a common disease found in 10% to 20% of cases having chronic watery diarrhea. Obvious endoscopically identifiable changes of the mucosal surface are usually absent, thus diagnosing microscopic colitis relies on multiple biopsy sampling from all segments of the colon. Chromoendoscopy using indigo-carmine dye spray might, however, unravel mucosal changes in microscopic colitis (Suzuki 2011).

The aim of this study is to investigate if chromoendoscopy using Indigo-Carmine 0.2-0.5% in patients with chronic watery diarrhea is useful in diagnosing microscopic colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic non-bloody diarrhea for at least one month

Exclusion Criteria:

* Patients who decline to participate
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Detection of microscopic colitis using chromoendoscopy | 12 month
  To investigate the usefullness of chromoendoscopy in diagnosing microscopic colitis using 0.2-0.5% Indigo-Carmine dye spray. The golden standard is the results of histological examination of biopsies from the colo-rectal mucosa.

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Schmidt, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karoliniska University Hospital, Dept. of Gastroenterology, Stockholm, Sweden

REFERENCES:
- [Background] Suzuki G, Mellander MR, Suzuki A, Rubio CA, Lambert R, Bjork J, Schmidt PT. Usefulness of colonoscopic examination with indigo carmine in diagnosing microscopic colitis. Endoscopy. 2011 Dec;43(12):1100-4. doi: 10.1055/s-0031-1291423. Epub 2011 Nov 4. PMID 22057822